CLINICAL TRIAL: NCT06990256
Title: Evaluation of Urolithin A and Fisetin on Improving Sleep and Aging Biomarkers in Middle-Aged and Older Adults: A Randomized Controlled Trial
Brief Title: Evaluation of Urolithin A and Fisetin on Improving Sleep and Aging Biomarkers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Wuhan Wuchang Hospital (Unknown); Abinopharm, Inc (Network)
Responsible Party: Principal Investigator, Liangkai Chen, Associate professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-008-01
Record Dates: First submitted 2025-05-09; First posted 2025-05-25 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-09

CONDITIONS: Sleep Disorder; Aging
Keywords: Urolithin A; Fisetin; Sleep Disorder; Aging
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Urolithin A Treatment Group (Experimental): Take a intervention capsule (containing 500 mg of Urolithin A) once daily after breakfast for a total of 12 weeks.
  Interventions: Dietary Supplement: Urolithin A intervention
- Fisetin Treatment Group (Experimental): Take a intervention capsule (containing 500 mg of Fisetin) once daily after breakfast for a total of 12 weeks.
  Interventions: Dietary Supplement: Fisetin intervention
- Combined Urolithin A and Fisetin Treatment Group (Experimental): Take a intervention capsule (containing 300 mg of Urolithin A + 200 mg of Fisetin) once daily after breakfast for a total of 12 weeks.
  Interventions: Dietary Supplement: Fisetin intervention; Dietary Supplement: Urolithin A intervention
- Placebo Control group (Placebo Comparator): Take a placebo capsule (containing 500 mg of corn starch) once daily after breakfast for a total of 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fisetin intervention — Participants assigned to this intervention take capsules containing a fixed dose of Fisetin daily after breakfast.
  Arms: Combined Urolithin A and Fisetin Treatment Group; Fisetin Treatment Group
Dietary Supplement: Placebo — Participants assigned to this intervention take a capsule containing 500 mg of corn starch daily after breakfast.
  Arms: Placebo Control group
Dietary Supplement: Urolithin A intervention — Participants assigned to this intervention take capsules containing a fixed dose of Urolithin A daily after breakfast.
  Arms: Combined Urolithin A and Fisetin Treatment Group; Urolithin A Treatment Group

SUMMARY:
The goal of this clinical trial is to evaluate the effects of Urolithin A (UA) and Fisetin on improving sleep and aging biomarkers in middle-aged and older adults. The main questions it aims to answer are:

Can UA and Fisetin improve sleep quality in middle-aged and older adults? Do these substances have a positive effect on aging biomarkers, such as inflammation, oxidative stress, and aging-related proteins? Researchers will compare four groups: Placebo group (a look-alike substance that contains no drug), 500 mg UA group, 500 mg Fisetin group and 300 mg UA + 200 mg Fisetin group.

Participants will:

Take the assigned capsules daily after breakfast for 12 weeks. Attend three clinic visits (baseline [Week 0], mid-intervention [Week 4], and post-intervention [Week 12]) including blood tests, sleep quality assessments (PSQI scale, actigraphy, polysomnography), and analysis of aging biomarkers (DNA methylation, inflammatory cytokines, etc.). Keep a sleep diary, complete a dietary survey, assess mental health, and measure frailty indicators. Provide stool and urine samples at baseline and post-intervention for gut microbiome and metabolite analysis. This trial aims to provide scientific evidence for the development of new nutritional intervention strategies to improve the healthy aging.

DETAILED DESCRIPTION:
The accelerating population aging has exacerbated the burden of chronic diseases among middle-aged and older adults, with sleep disorders emerging as a core health issue that forms a vicious cycle with aging. Urolithin A and Fisetin as dietary bioactive components have gained attention for their potential health benefits, including anti-aging, anti-inflammatory, and antioxidant properties. However, researches on their effects in sleep and aging remain limited, and clinical evidence for their combined intervention is currently lacking. This study aims to evaluate the effects of Urolithin A and Fisetin on improving sleep and aging biomarkers in middle-aged and older adults, providing scientific evidence for developing new scientific dietary strategies. It is a randomized controlled trial. A total of 80 participants will be recruited and randomly assigned to four groups: control group, Urolithin A 500 mg group, Fisetin 500 mg group, and Urolithin A 300 mg + Fisetin 200 mg group. The intervention period will last 12 weeks, with all participants taking one capsule of the intervention substance or placebo daily after breakfast. Primary outcomes include subjective and objective sleep quality assessments and frailty assessment. Secondary outcomes include metabolic, immune and inflammatory markers, gut microbiota analysis and quality of life assessment. Participants will undergo three follow-up assessments: baseline (week 0), mid-intervention (week 4), and end of intervention (week 12). Data will be analyzed using SAS 9.4 following the intention-to-treat principle. It is expected to provide preliminary data on the single and combined effects of Urolithin A and Fisetin on improving sleep and aging biomarkers in middle-aged and older adults, as well as reveal their potential synergistic effects. The rigorous and innovative design will serve as a reference for future mechanistic studies, which has important public health significance.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30-75 years;
* Total score > 5 points on the Pittsburgh Sleep Quality Index (PSQI) for sleep quality assessment;
* Able to use personal mobile devices for WeChat, internet access, and related operations;
* Informed about the intervention trial and willing to undergo sleep monitoring and other examinations during the study;
* Commitment to consume coffee, strong tea, or alcohol ≤1 time per week during the trial period;

Exclusion Criteria:

* Participation in any clinical trials or dietary/exercise intervention programs within the past 3 months or concurrently;
* Diagnosis of major mental disorders or family history thereof, or current use of psychotropic drugs or mood-regulating medications;
* Experiencing major psychological trauma (e.g., death of a close relative, significant financial loss) personally or within the family in the past 3 months;
* Severe diseases affecting inflammatory levels and/or endocrine components (e.g., severe obesity, uncontrolled diabetes or poorly controlled blood glucose, myocardial infarction, cerebral infarction);
* Current use of hormonal medications, beta-blockers, steroids, non-steroidal anti-inflammatory drugs (NSAIDs), etc.;
* Use of medications potentially affecting sleep or aging biomarkers (e.g., melatonin, antidepressants, anxiolytics) within the past 3 months;
* Plans for relocation or long-term travel within the next 6 months, which may hinder continuous intervention and follow-up.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Subjective Sleep Quality Score | From enrollment to the end of intervention at 12 weeks
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI), developed by psychiatrist Dr. Buysse in 1989. The PSQI includes seven components: subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbance, used sleep medication, and daytime dysfunction. Each component score ranges from 0 to 3, with a total score ranges from 0 to 21. Higher scores indicate poorer sleep quality, and a total score >7 suggests clinically significant sleep impairment.
Chronotype | From enrollment to the end of intervention at 12 weeks
  Chronotype will be evaluated using the Morningness-Eveningness Questionnaire (MEQ), a self-reported scale consisting of 19 items assessing physiological and behavioral preferences across a 24-hour cycle. MEQ-5 will be used in this trial, which scores range from 4 to 25, with higher scores indicating a morning-oriented chronotype and lower scores reflecting an evening-oriented preference.
Polysomnography | From enrollment to the end of intervention at 12 weeks
  Polysomnography (PSG) is a comprehensive sleep assessment and the reference standard for objectively evaluating sleep physiology and sleep disorders. It records multiple signals during sleep, typically including electroencephalography, electrooculography, and electromyography, as well as respiratory airflow and effort, oxygen saturation, electrocardiography, and body position/limb movements, to characterize sleep stages, sleep architecture, and sleep-related events. PSG is commonly used to assess sleep-disordered breathing (e.g., obstructive sleep apnea), periodic limb movement disorder, and REM sleep behavior disorder. All PSG data in this study will be scored and analyzed according to American Academy of Sleep Medicine (AASM) guidelines.

SECONDARY OUTCOMES:
Number of participants with abnormal blood and urine routine tests results | From enrollment to the end of intervention at 12 weeks
  We will conduct blood routine and urine routine tests, and report the number of people with abnormal tests results. The tests indicators include: Red Blood Cell Count (RBC), Hemoglobin (Hb), Hematocrit (Hct), White Blood Cell Count (WBC), Neutrophils (Neut# and Neut%), Lymphocytes (Lym# and Lym%), Monocytes (Mono# and Mono%), Platelet Count (PLT), Mean Corpuscular Volume (MCV), Mean Corpuscular Hemoglobin (MCH), Mean Corpuscular Hemoglobin Concentration (MCHC), Urine Physical Characteristics (Appearance, specific gravity, pH), Urine Biochemical Analysis (Protein, Glucose, Occult blood, Leukocytes, Erythrocytes, and Bacteria). Any abnormal results will be marked on the laboratory report.
Homeostatic Model Assessment of Insulin Resistance | From enrollment to the end of intervention at 12 weeks
  Plasma samples collected at different time points will be classified and labeled with two sets of each sample. An automated hematology analyzer in the hospital will be used.The degree of Insulin Resistance (IR) and sensitivity will be calculated by the Homeostatic Model Assessment (HOMA-IR) using the formula:
  HOMA-IR=(Fasting Insulin (μIU/mL) × Fasting Glucose (mmol/L) )/22.5
Frailty Assessment | From enrollment to the end of intervention at 12 weeks
  Frailty status will be evaluated using the Fried Frailty Phenotype. The Fried Frailty Phenotype includes exhaustion, weight loss, low physical activity, slow gait speed, and grip strength measurement.For consistency with previous literature, participants who meet 3 or more criteria will be diagnosed as frailty, those who meet 1 or 2 criteria will be classified as prefrailty, and those who meet none of the criteria will be considered as nonfrailty.
Fatigue Severity Scale Score | From enrollment to the end of intervention at 12 weeks
  The Fatigue Severity Scale will be used to measure the fatigue score of participants.Evaluates fatigue severity over the past week through 9 items, with each item scored from 1 (strongly disagree) to 7 (strongly agree). The total score ranges from 9 to 63. Higher scores indicate more severe fatigue.
Patient Health Questionnaire-9 Score | From enrollment to the end of intervention at 12 weeks
  The Patient Health Questionnaire-9 (PHQ-9) is a brief self-report scale commonly used in clinical practice to assess depressive symptoms. It consists of 9 questions, primarily asking about the experience of depressive symptoms over the past two weeks and their frequency. Each response is set from 0 (not at all) to 3 (nearly every day), with a total score range of 0 to 27. Higher scores indicate more severe depressive symptoms.
Generalized Anxiety Disorder Scale Score | From enrollment to the end of intervention at 12 weeks
  The Generalized Anxiety Disorder Scale (GAD-7) is a brief self-report scale used to assess anxiety symptoms over the past two weeks. It includes 7 questions, with responses rated from 0 to 3. The total score ranges from 0 to 21. Higher scores indicate more severe anxiety symptoms.
Determination of Plasma Immunoglobulin Levels (g/L) | From enrollment to the end of intervention at 12 weeks
  The levels of immunoglobulin A (IgA), immunoglobulin G (IgG), and immunoglobulin M (IgM) in plasma samples will be measured using a fully automated biochemical analyzer, with all units expressed as g/L.
DNA Methylation Clock | From enrollment to the end of intervention at 12 weeks
  The DNA methylation clock is an algorithm that integrates DNA methylation measurements across the genome to quantify biological age changes. It is considered a highly accurate molecular marker of human biological age. This clock can detect DNA methylation age reversal up to three months in advance, thus showing potential for quantifying biological aging, assessing expected lifespan, or evaluating the efficacy of interventions.
Profile of Mood States-Short Form (Chinese Version) Score | From enrollment to the end of intervention at 12 weeks
  The Profile of Mood States-Short Form (Chinese Version) will be used to measure the energy score of participants. It measures energy levels using a 5-point scale ranging from 0 (never) to 4 (extremely), total score ranges from 0 to 160. Higher scores indicate greater vitality.
Plasma Interleukin Levels | From enrollment to the end of intervention at 12 weeks
  Plasma interleukin levels are primarily used to reflect the inflammatory and immune status. In this study, the concentrations of interleukins (IL-1β, IL-6, IL-8, IL-10, IL-11, IL-33, IL-23R, and IL-17A) will be measured in fasting plasma samples of participants using ELISA kits, with units expressed as pg/mL. Notably, IL-11, IL-33, IL-23R, and IL-17A have recently gained attention as key molecules associated with aging.
Gut Microbiota Diversity Analysis (Based on 16S rRNA Gene Sequencing) | From enrollment to the end of intervention at 12 weeks
  Stool samples (10g) from participants will be collected. These samples will be rapidly frozen in dry ice to stop metabolic reactions. DNA will be extracted from the frozen stool samples using the GNOME DNA isolation kit, and 16S rRNA sequencing will be performed using the IlluminaHiSeq2500 platform. 16S rRNA gene sequencing is a common method for analyzing the composition of the gut microbiota by high-throughput sequencing technology, widely used to assess the diversity and structural changes of the gut microbiota. The process includes DNA extraction from stool samples, amplification of specific regions of the 16S rRNA gene (such as the V3-V4 regions), and sequencing of the amplicons using a high-throughput sequencing platform (e.g., Illumina). Data quality control and microbiome structure analysis will be performed using bioinformatics tools (such as QIIME, Mothur and USEARCH) to assessing diversity.
D-lactic acid level | From enrollment to the end of intervention at 12 weeks
  D-lactic acid level (μmol/L) in peripheral blood will be measured as an indicator of intestinal mucosal barrier integrity. Under physiological conditions, circulating D-lactic acid remains at trace concentrations in micromolar range. Elevated serum level reflects increased intestinal permeability due to mucosal damage from inflammation or ischemia, allowing bacterial-derived D-lactic acid to enter circulation.
NAD+ Level Measurement | From enrollment to the end of intervention at 12 weeks
  Nicotinamide adenine dinucleotide (NAD+) plays a crucial role in cellular energy metabolism, redox reactions, and aging, which will be evaluated to monitor metabolic status and intervention efficacy. Methods include high-performance liquid chromatography (HPLC), mass spectrometry (MS), HPLC-MS/MS, and ELISA. Although ELISA has relatively lower accuracy, it is convenient to use. For this study commercial ELISA kits will be used.
Quality of Life Assessment | From enrollment to the end of intervention at 12 weeks
  The World Health Organization Quality of Life Brief Version (WHOQOL-BREF) will be administered at baseline (week 0) and the end of intervention (week 12) to assess changes across four domains: physical health, psychological status, social relationships, and environmental factors. This instrument assesses the overall impact of the intervention on participants' quality of life.The standardized scores range from 0 to 100, with higher scores indicating a better quality of life.
Arterial stiffness assessment | From enrollment to the end of intervention at 12 weeks
  Arterial stiffness will be assessed as a secondary outcome using an automated, noninvasive oscillometric vascular screening system. Bilateral brachial and ankle blood pressures and pulse waveforms will be recorded to derive brachial-ankle pulse wave velocity (baPWV) and the ankle-brachial index (ABI), along with peripheral blood pressure and heart rate, following standardized resting conditions and the manufacturer's recommended procedures.
Cardiopulmonary exercise testing | From enrollment to the end of intervention at 12 weeks
  Cardiopulmonary exercise testing (CPET) will be conducted using an incremental, symptom-limited protocol on an electronically braked cycle ergometer. Participants will complete standardized pre-test screening and resting measurements, followed by a brief warm-up and stepwise increases in workload until volitional exhaustion or predefined termination criteria are met. Breath-by-breath gas exchange will be measured continuously to derive oxygen uptake (VO₂), carbon dioxide production (VCO₂), and minute ventilation (VE), alongside concurrent monitoring of heart rate, blood pressure, and electrocardiography. Key outcomes will include peak oxygen uptake (VO₂peak) and ventilatory threshold-based indices, with test procedures and interpretation aligned with established CPET guidelines.

CONTACTS AND LOCATIONS:
Locations (1):
- Wuchang Hospital Affiliated to Wuhan University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No